CLINICAL TRIAL: NCT05436379
Title: Treatment, Emotion, and Neuromodulation of Depression (TREND) Study
Acronym: TREND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erika Forbes (Other)
Responsible Party: Sponsor-Investigator, Erika Forbes, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21060041
Record Dates: First submitted 2022-02-04; First posted 2022-06-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Positive Affect; Theta Burst Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The proposed study will use theta burst stimulation (TBS) in an open-label, non-randomized open study for young adults with depression. The study will include measurement of brain function before and after TBS to investigate treatment mechanisms. A subset of participants will also complete a training to enhance positive emotions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TBS (Other): In this open-label trial, all participants will undergo 2 or 3 continuous TBS (cTBS) sessions per visit over 10 days (weekdays, over 2 weeks; total = 20 or 30 TBS sessions in 10 visits). The total time of each pair of sessions (including pause between sessions) will be approximately 1 hour, with each session lasting approximately 100 seconds.
  There is only 1 group and 1 arm of the study. All participants will receive the treatment.
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — TBS, a next-gen form of transcranial magnetic stimulation (TMS), requires shorter duration and frequency of stimulation and provides comparable clinical efficacy to traditional repetitive TMS for depression. Thus it is an appropriate technique for use with young adults with depression. TBS can be delivered safely and effectively on an accelerated schedule with two sessions/day. Based on an earlier (ongoing) study of TBS to dorsomedial prefrontal cortex, investigators will administer TBS to dmPFC over 2 weeks in young adults with depression. Addressing the behavioral aspects of anhedonia and reward processing, a subset of participants will also receive positive affect training. Magnetic resonance imaging will guide the personalized location of TBS and will be used to examine change in frontostriatal circuitry with TBS. This study has the potential to influence development of new treatments for depression and anhedonia, with possible mechanisms in frontostriatal brain function.

SUMMARY:
The investigators will administer theta burst stimulation (TBS) in efforts to observe a decrease in severity of reported depression symptoms. A subset of participants will receive positive affect training during this intervention.

DETAILED DESCRIPTION:
The study has a longitudinal design in which participants complete a baseline assessment, 20 or 30 theta burst stimulation (TBS) sessions, a post-TBS assessment, and a follow-up assessment 4 months later. Ideally, TBS sessions will be delivered two or three times a day, 5 days/week, for 2 weeks. This procedural design of a shorter treatment duration is based on findings of pattern of improvement and newly developed SAINT protocol. A subset of participants will receive training in enhancing positive affect, with 10 training sessions occurring between pairs of TBS sessions. In this study, "response" to intervention will be defined as a greater than 50% decrease in severity of depression symptoms reported by participants.

ELIGIBILITY:
Inclusion Criteria:

* Current Diagnostic and Statistical Manual (DSM-5) Depressive Disorder

Exclusion Criteria:

* Bipolar disorder (lifetime)
* Obsessive-compulsive disorder (lifetime)
* History of psychosis
* Daily use of nicotine
* Past-month use of cocaine, amphetamines, Methyl enedioxy methamphetamine (MDMA), Phencyclidine (PCP), Ketamine, or gamma-hydroxybutyrate (GHB)
* Past 6 month substance use disorder
* Binge drinking (using NIAAA criteria) within the past week, alcohol use in the past 12 hours
* Neurological disorders: Epilepsy, Parkinson's Disease, brain tumor, brain injury, stroke
* History of head trauma with a loss of consciousness (e.g., concussion)
* History of seizures
* MRI contraindications: body shape/size too large to fit in scanner, claustrophobia, and ferromagnetic metal in the body
* Pregnancy
* Current use of Clozapine, Bupropion, or prescription stimulants
* Current use of benzodiazepines or mood stabilizers
* Body shape/size too large to fit in MRI scanner
* Claustrophobia
* Metal in the head or ferromagnetic metal in the rest of the body
* Implanted medical devices
* High-risk suicidality

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
depression severity | up to 1 year
  Score on the Montgomery-Asberg Depression Rating Scale (MADRS), administered by a study team member

CONTACTS AND LOCATIONS:
Overall Officials: Erika E Forbes, Ph.D, Principal Investigator — University of Pittsburgh
Locations (1):
- The University of Pittsburgh, Department of Psychiatry, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Der-Avakian A, Markou A. The neurobiology of anhedonia and other reward-related deficits. Trends Neurosci. 2012 Jan;35(1):68-77. doi: 10.1016/j.tins.2011.11.005. Epub 2011 Dec 15. PMID 22177980
- [Background] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Background] Dunlop K, Gaprielian P, Blumberger D, Daskalakis ZJ, Kennedy SH, Giacobbe P, Downar J. MRI-guided dmPFC-rTMS as a Treatment for Treatment-resistant Major Depressive Disorder. J Vis Exp. 2015 Aug 11;(102):e53129. doi: 10.3791/53129. PMID 26327307
- [Background] Forbes EE. Where's the fun in that? Broadening the focus on reward function in depression. Biol Psychiatry. 2009 Aug 1;66(3):199-200. doi: 10.1016/j.biopsych.2009.05.001. No abstract available. PMID 19577042
- [Background] Healey KL, Morgan J, Musselman SC, Olino TM, Forbes EE. Social anhedonia and medial prefrontal response to mutual liking in late adolescents. Brain Cogn. 2014 Aug;89:39-50. doi: 10.1016/j.bandc.2013.12.004. Epub 2014 Jan 10. PMID 24412087
- [Background] Kessler RC, Rose S, Koenen KC, Karam EG, Stang PE, Stein DJ, Heeringa SG, Hill ED, Liberzon I, McLaughlin KA, McLean SA, Pennell BE, Petukhova M, Rosellini AJ, Ruscio AM, Shahly V, Shalev AY, Silove D, Zaslavsky AM, Angermeyer MC, Bromet EJ, de Almeida JM, de Girolamo G, de Jonge P, Demyttenaere K, Florescu SE, Gureje O, Haro JM, Hinkov H, Kawakami N, Kovess-Masfety V, Lee S, Medina-Mora ME, Murphy SD, Navarro-Mateu F, Piazza M, Posada-Villa J, Scott K, Torres Y, Carmen Viana M. How well can post-traumatic stress disorder be predicted from pre-trauma risk factors? An exploratory study in the WHO World Mental Health Surveys. World Psychiatry. 2014 Oct;13(3):265-74. doi: 10.1002/wps.20150. PMID 25273300
- [Background] Morgan JK, Shaw DS, Olino TM, Musselman SC, Kurapati NT, Forbes EE. History of Depression and Frontostriatal Connectivity During Reward Processing in Late Adolescent Boys. J Clin Child Adolesc Psychol. 2016;45(1):59-68. doi: 10.1080/15374416.2015.1030753. Epub 2015 Apr 27. PMID 25915469
- [Background] Romens SE, Casement MD, McAloon R, Keenan K, Hipwell AE, Guyer AE, Forbes EE. Adolescent girls' neural response to reward mediates the relation between childhood financial disadvantage and depression. J Child Psychol Psychiatry. 2015 Nov;56(11):1177-84. doi: 10.1111/jcpp.12410. Epub 2015 Apr 5. PMID 25846746
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650